CLINICAL TRIAL: NCT03915808
Title: The Effects of Supplementation of Conjugated Linoleic Acid on Body Fat Reduction in Overweight or Obesity Chinese Adults During Weight Loss: A Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: The Effects of Supplementation of Conjugated Linoleic Acid on Body Fat Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jiaomei Yang (Other)
Responsible Party: Sponsor-Investigator, Jiaomei Yang, Associate Research Fellow, Xi'an Jiaotong University
Organization: Xi'an Jiaotong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20190201
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This will be a parallel randomized, double-blinded, placebo-controlled trial. Sixty-six overweight or obese men and women aged from 18 to 50 years with elevated body fat percentage, who also meet our inclusion and exclusion criteria, will be randomly assigned to: the treatment group, daily supplementation of 3.2 g CLA (Cis-9, trans-11 isomers and trans-10, cis-12 isomers) plus lifestyle counselling weight loss program; or the control group, daily supplementation of sunflower oil. The intervention will include a 3-day run-in phase and 12-week interventional phase. At baseline and the end of the intervention, physical examination including questionnaires, anthropometric measurement, body composition by Dual Energy X-ray Absorptiometry (DXA), biological sample collection will be undertaken. During the invention, regular lifestyle counselling sessions will be delivered, and detailed record will be tracked for all participants to monitor and improve the adherence and safety.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conjugated linoleic acid plus lifestyle counselling (Experimental): supplementation of 3.2 g/day conjugated linoleic acid and receive education sessions regularly
  Interventions: Dietary Supplement: Conjugated linoleic acid group
- Sunflower oil plus lifestyle counselling (Placebo Comparator): supplementation of equivalent sunflower oil, and receive education sessions regularly
  Interventions: Dietary Supplement: Sunflower oil group

INTERVENTIONS:
Dietary Supplement: Conjugated linoleic acid group — supplementation of 3.2 g/day conjugated linoleic acid in 8 capsules, and receive education sessions every four weeks (Dietary and lifestyle counselling, featured with low fat and low added sugar, moderate physical activity)
  Arms: Conjugated linoleic acid plus lifestyle counselling
Dietary Supplement: Sunflower oil group — supplementation of equivalent sunflower oil in 8 capsules, and receive education sessions every four weeks (Dietary and lifestyle counselling, featured with low fat and low added sugar, moderate physical activity)
  Arms: Sunflower oil plus lifestyle counselling

SUMMARY:
This is a double-blinded randomized controlled trial, to evaluate the effectiveness of daily supplementation of 3.2 g CLA on body fat reduction and lipid profile in overweight or obese Chinese adults, during a lifestyle counselling-based weight loss.

DETAILED DESCRIPTION:
This will be a parallel randomized, double-blinded, placebo-controlled trial. Sixty-six overweight or obese men and women aged from 18 to 45 years with elevated body fat percentage, who also meet our inclusion and exclusion criteria, will be randomly assigned to: the treatment group, daily supplementation of 3.2 g CLA (Cis-9, trans-11 isomers and trans-10, cis-12 isomers) plus lifestyle counselling weight loss program; or the control group, daily supplementation of sunflower oil. The intervention will include a 3-day run-in phase and 12-week interventional phase. At baseline and the end of the intervention, physical examination including questionnaires, anthropometric measurement, body composition by Dual Energy X-ray Absorptiometry (DXA), biological sample collection will be undertaken. During the invention, regular lifestyle counselling sessions will be delivered, and detailed record will be tracked for all participants to monitor and improve the adherence and safety.

ELIGIBILITY:
Inclusion Criteria:

1) Body fat percentage ≥ 20% for men, Body fat percentage ≥ 30% for women ; 2) aged from 18 to 45 years old.

Exclusion Criteria:

1. Pregnancy or lactation;
2. Abnormal liver or kidney function indicated by physical examination within 6 months;
3. Gastrointestinal problems that affect the complying with the procedure;
4. Sever cardiovascular disease;
5. Active cancer;
6. Mental diseases, epilepsy or using anti-depression drugs;
7. Using medicine that affect body weight;
8. Participating in other scientific studies within 3 months before the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-07-21 (Actual)

PRIMARY OUTCOMES:
Change of body fat percentage | week 0 and week 12

SECONDARY OUTCOMES:
Change of body fat mass | week 0 and week 12
Change of body mass index | week 0 and week 12
Change of weight | week 0, week 4, week 8, and week 12
Change of waist circumference | week 0 and week 12
Change of triglycerides | week 0 and week 12
Change of total cholesterol | week 0 and week 12
Change of LDL-cholesterol | week 0 and week 12
Change of HDL-cholesterol | week 0 and week 12
Change of blood pressure | week 0 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Xin Liu, PhD, Principal Investigator — Xi'an Jiaotong University Health Science Center
Locations (1):
- Xi'an Jiaotong University Health Science Center, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jia K, She Y, He Y, He J, He Y, Xu K, Ma G, Li W, He C, Feng X, Wang M, Tang A, Sun X, Kong L, Liu X. Conjugated Linoleic Acid Supplementation Suppresses the De Novo Lipogenesis in Adults With High Body Fat: A Double-Blind, Randomized, Placebo-Controlled Trial. Mol Nutr Food Res. 2025 Dec;69(24):e70306. doi: 10.1002/mnfr.70306. Epub 2025 Oct 30. PMID 41169023
- [Derived] He Y, Xu K, Li Y, Chang H, Liao X, Yu H, Tian T, Li C, Shen Y, Wu Q, Liu X, Shi L. Metabolomic Changes Upon Conjugated Linoleic Acid Supplementation and Predictions of Body Composition Responsiveness. J Clin Endocrinol Metab. 2022 Aug 18;107(9):2606-2615. doi: 10.1210/clinem/dgac367. PMID 35704027
- [Derived] Chang H, Gan W, Liao X, Wei J, Lu M, Chen H, Wang S, Ma Y, Wu Q, Yu Y, Liu X. Conjugated linoleic acid supplements preserve muscle in high-body-fat adults: A double-blind, randomized, placebo trial. Nutr Metab Cardiovasc Dis. 2020 Sep 24;30(10):1777-1784. doi: 10.1016/j.numecd.2020.05.029. Epub 2020 Jun 8. PMID 32684362